CLINICAL TRIAL: NCT05516485
Title: Measuring Brain Tumor Consistency Using Magnetic Resonance Elastography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6B-20-2; NCI-2021-05851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6B-20-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-08-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Restraint, Physical; Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (MRE, tumor grading) (Experimental): Patients undergo MRE scan over 25 minutes before surgery at the time of standard of care pre-operative MRI scan. On the day of surgery, the surgeon grades and records tumor consistency/stiffness during the operation and afterwards.
  Interventions: Other: Assessment; Device: Magnetic Resonance Elastography

INTERVENTIONS:
Other: Assessment — Undergo grading and recording of tumor consistency/stiffness
  Other Names: Assess
Device: Magnetic Resonance Elastography — Undergo MRE
  Other Names: MRE

SUMMARY:
This clinical trial tests whether a new imaging technique called magnetic resonance elastography (MRE) is useful in determining the consistency of brain tumors and whether this could be used to guide surgical planning and choice of approach (the type of surgery that is needed) for patients with brain tumors. Comparing MRE with the typical magnetic resonance imaging (MRI) scan may help researchers assess the quality, reliability, and diagnostic utility of this scan when evaluating brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine tolerance interval of MRE measurement in kilopascals (kPa) and associated distribution of percent stiff (hard) and soft tumors above the higher limit and below the lower limit.

II. Through machine learning with MRE and clinical/demographic factors, to identify diagnostic thresholds in separating stiff tumor from soft tumor.

OUTLINE:

Patients undergo MRE scan over 25 minutes before surgery at the time of standard of care pre-operative MRI scan. On the day of surgery, the surgeon grades and records tumor consistency/stiffness during the operation and afterwards.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older who undergo surgical resection for brain tumor at Keck Medical Center of University of South Carolina (USC) are eligible for inclusion into this study

Exclusion Criteria:

* Patients who cannot tolerate MRE
* Those ineligible for MRI due to metallic implants, claustrophobia, or body habitus too large to fit in our MRI machine
* Those not undergoing surgical resection of brain tumor
* Children under the age of 18, pregnant women, wards of the state, and prisoners
* There will be no exclusion of patients based on gender, racial or ethnic origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Tumor stiffness (hardness) (based on surgeon's grading) | Baseline to 6 weeks
  Surgeon will grade tumor stiffness based on the Zada scale of 1-5, with stiffer tumors receiving higher scores on the scale, as follows: 1) extremely soft tumor, internal debulking with suction only; 2) soft tumor, internal debulking mostly with suction, and remaining fibrous strands resected with easily folded capsule; 3) average consistency, tumor cannot be freely suctioned and requires mechanical debulking, and the capsule then folds with relative ease; 4) firm tumor, high degree of mechanical debulking required, and capsule remains difficult to fold; and 5) extremely firm, calcified tumor, approaches density of bone, and capsule does not fold. Outcome will be further dichotomized into two categories: soft (1, 2) vs. stiff (hard).
Tumor stiffness (based on MRE) | Baseline to 6 weeks
  The tumor stiffness as measured by MRE in kilopascals (kPa) will be analyzed to establish 2 cut-points. (1) Higher cut-point: Because higher kPa is a quality of stiffer (harder) tumors the high cut off point will be the kPa at which no tumor greater than or equal to that value can be called soft. (2) Lower cut-point: this will be the kPa at which no tumor lower than or equal to that value can be called stiff (hard).

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Shiroishi, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States